CLINICAL TRIAL: NCT03473561
Title: Efficacy and Safety of Racecadotril in the Treatment of Taiwanese Children Aged 3 to 60 Months Suffering From Acute Diarrhea: A Prospective, Open-label, Multicenter, Single-arm Study.
Brief Title: Study to Evaluate the Efficacy and Safety of Racecadotril in Children Aged 3 to 60 Months Suffering From Acute Diarrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RACE3002
Record Dates: First submitted 2018-03-12; First posted 2018-03-22 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-02

CONDITIONS: Diarrhea, Infantile
MeSH Terms: conditions — Diarrhea, Infantile | interventions — racecadotril; ORALIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Racecadotril plus standard treatment oral rehydration solution (Experimental): Racecadotril Infants Granules for Oral Suspension 10 mg (in addition to standard treatment i.e. oral rehydration solution) Racecadotril Children Granules for Oral Suspension 30 mg (in addition to standard treatment i.e. oral rehydration solution)
  Interventions: Drug: Racecadotril plus ORS

INTERVENTIONS:
Drug: Racecadotril plus ORS — 1.5 mg/kg of Racecadotril will be administered, 3 times daily, via the oral route (in addition to standard treatment i.e. oral rehydration solution).
  In infants less than 9 kg: one 10 mg sachet 3 times daily. In infants from 9 kg to < 13 kg: two 10 mg sachets 3 times daily. In children from 13 kg to 27 kg: one 30 mg sachet 3 times daily. In children of more than 27 kg: two 30 mg sachets 3 times daily.

SUMMARY:
This is a prospective, open-label, multicenter, single-arm study evaluating the efficacy and safety of Racecadotril the treatment of children aged 3 to 60 months suffering from acute diarrhea

DETAILED DESCRIPTION:
Subjects presenting with acute diarrhea will be evaluated for eligibility. If eligible, demographics, number of stools during the last 12 hours will be assessed as baseline values. On Day 1, the subject will start with study treatment.

Subjects will be treated with Racecadotril three times daily according to the body weight dose requirement on an out-patient basis for maximum 5 days in addition to ORS. ORS will be prescribed by the investigator. The parent(s)/caregiver(s)/legal representative(s) will be instructed to stop treatment when the patient recovered. Recovery is defined by the evacuation of the first of two consecutive normal stools or no stool within 12 hours. In the evening of each day, the parent(s)/caregiver(s)/legal representative(s) will fill in their diaries, documenting date and time of each individual stool, the stool consistency of each stool, ORS amount and the study drug intake. AEs are to be reported on an ongoing basis.

The last dose of study drug intake will be the morning dose of day 6, if not recovered earlier. The parent(s)/caregiver(s)/legal representative(s) will visit the site for the end of study visit of the child. Data on vital signs, AEs, physical examination and concomitant medication will be collected. The parent(s)/caregiver(s)/legal representative(s) will return the diaries and unused medication.

A phone call contact will be performed 5-7 days after the end of the treatment period or recovery for the safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from one of the parent(s)/legal representative(s)
* Subjects, both genders, aged 3 to 60 months
* Subjects with acute diarrhea (defined as the passage of three or more unformed or liquid stools within the last 24 hours and lasting for less than 3 days)

Exclusion Criteria:

* Known allergy to Racecadotril or any of its ingredients
* Subjects suffering from renal or hepatic impairment
* Subjects with fever > 39 degrees Celsius
* Subjects with bloody and/or purulent stools
* Subjects suffering from antibiotic (e.g. amoxicillin)-associated diarrhea, chronic diarrhea or iatrogenic diarrhea
* Subjects with alternating bouts of diarrhea and constipation
* Diarrhea due to exacerbation of chronic gastrointestinal diseases such as irritable bowel syndrome, irritable bowel disease or pancreatic exocrine insufficiency
* Cystic fibrosis or coeliac disease
* Subjects suffering from prolonged or uncontrolled vomiting
* Subjects with rare hereditary problems of fructose intolerance, glucose-galactose malabsorption syndrome or sucrase isomaltase insufficiency
* Subjects having received antibiotic treatment at any time within 2 weeks prior to inclusion into the study
* Subjects having received antidiarrheal drugs 48 hours prior to inclusion into the study
* Subjects with severe dehydration requiring intravenous fluid, electrolyte replacement or hospitalization treatment
* Subject with a history of angioedema or who had reported angioedema with angiotensin converting enzyme inhibitors (such as captopril, enalapril, lisinopril, perindopril, ramipril)
* Subjects with combined diseases or medical situations that would prevent to be enrolled into the study, depending on the judgment of the investigator
* Intake of experimental drug within 30 days prior to study start
* Subjects with contraindications to ORS or susceptible to the warnings of ORS

Ages: 3 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2018-08-25 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Linkou Chang Gung Memorial Hospital, Taipei
  - Mackay Memorial Hospital, Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- Racecadotril Plus Standard Treatment Oral Rehydration Solution: Racecadotril Infants Granules for Oral Suspension 10 mg (in addition to standard treatment i.e. oral rehydration solution) Racecadotril Children Granules for Oral Suspension 30 mg (in addition to standard treatment i.e. oral rehydration solution)
  Racecadotril plus ORS: 1.5 mg/kg of Racecadotril will be administered, 3 times daily, via the oral route (in addition to standard treatment i.e. oral rehydration solution).
  In infants less than 9 kg: one 10 mg sachet 3 times daily. In infants from 9 kg to < 13 kg: two 10 mg sachets 3 times daily. In children from 13 kg to 27 kg: one 30 mg sachet 3 times daily. In children of more than 27 kg: two 30 mg sachets 3 times daily.
Period: Overall Study
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: FA sample
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 31
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 31

OUTCOME MEASURES:

1. Primary Outcome: Duration of Diarrhea (Hours) Between the Start of Treatment Until Last Diarrheal/Watery Stool Before Recovery or End of Study Treatment (Treatment Duration Maximal 5 Days
Description: Duration of diarrhea is defined by date and time of the evacuation of the final diarrheal stool derived from the daily diary
Time Frame: 5 days
Measure: Mean (Standard Error); unit: hours
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution
Number analyzed (Participants) | 31
hours | 57.5 (5.79)

2. Secondary Outcome: Number of Recovered Subjects
Description: Number of recovered subjects
Time Frame: 5 days
Population: FA Sample
Measure: Count of Participants; unit: Participants
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution
Number analyzed (Participants) | 31
Participants | 23

3. Secondary Outcome: Global Physician Assessment at the End of Treatment
Description: Scores 1-6 (Scores 1 and 2 are defined as success)
Time Frame: 5 days
Measure: Count of Participants; unit: Participants
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution
Number analyzed (Participants) | 31
Participants | 25

ADVERSE EVENTS:
Time Frame: 5 days plus 1 gap day
Arm/Group | Racecadotril Plus Standard Treatment Oral Rehydration Solution
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 16/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Racecadotril Plus Standard Treatment Oral Rehydration Solution (N=31)
Bronchitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Racecadotril Plus Standard Treatment Oral Rehydration Solution (N=31)
Diarrhoea (Gastrointestinal disorders) | 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 7
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 2
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT03473561/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT03473561/SAP_001.pdf